CLINICAL TRIAL: NCT02390037
Title: Pipeline™ Flex Embolization Device With Shield Technology™ Clinical Study
Acronym: PFLEX
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: NV PED 09
Record Dates: First submitted 2015-03-06; First posted 2015-03-17 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The objective of the study is to assess the incidence of safety outcomes in patients treated with Pipeline™ Flex embolization device with Shield Technology™.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent using the IRB/EC-approved consent form and agrees to comply with protocol requirements.
2. Age 18-80 years.
3. Subject has already been selected for flow diversion therapy as the appropriate treatment.
4. Subject has an unruptured target intracranial aneurysm (IA).
5. Subject has a target IA located in the anterior or posterior circulation.

Exclusion Criteria:

1. Major surgery in the past 30 days.
2. Any known contraindication to treatment with the Pipeline™ Flex embolization device with Shield Technology™ per Instructions for Use.
3. Pregnant or breast-feeding women or women who wish to become pregnant during the length of study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neuroradiologists and surgeons practice
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-03; Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of major stroke or neurological death | 1 year

SECONDARY OUTCOMES:
Device related neurologic adverse event rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Boccardi, M.D., Principal Investigator — Ospedale Niguarda "Ca' Granda"
Locations (7):
- Ziekenhuis Oost-Limburg, Genk, Belgium
- Germany (2):
  - Uniklinik Koln, Cologne
  - Alfried Krupp Krankenhaus, Essen
- Hellenic Air Force Hospital, Athens, Greece
- IRCCS Fondazione Istituto Neurologico C Besta, Milan, Italy
- Hospital Clinico Universitario de Valladolid, Valladolid, Spain
- Queen Elizabeth Hospital Birmingham, Birmingham, United Kingdom

REFERENCES:
- [Derived] Martinez-Galdamez M, Lamin SM, Lagios KG, Liebig T, Ciceri EF, Chapot R, Stockx L, Chavda S, Kabbasch C, Farago G, Nordmeyer H, Boulanger T, Piano M, Boccardi EP. Treatment of intracranial aneurysms using the pipeline flex embolization device with shield technology: angiographic and safety outcomes at 1-year follow-up. J Neurointerv Surg. 2019 Apr;11(4):396-399. doi: 10.1136/neurintsurg-2018-014204. Epub 2018 Sep 27. PMID 30262655
- [Derived] Martinez-Galdamez M, Lamin SM, Lagios KG, Liebig T, Ciceri EF, Chapot R, Stockx L, Chavda S, Kabbasch C, Farago G, Nordmeyer H, Boulanger T, Piano M, Boccardi EP. Periprocedural outcomes and early safety with the use of the Pipeline Flex Embolization Device with Shield Technology for unruptured intracranial aneurysms: preliminary results from a prospective clinical study. J Neurointerv Surg. 2017 Aug;9(8):772-776. doi: 10.1136/neurintsurg-2016-012896. Epub 2017 Feb 20. PMID 28223428